CLINICAL TRIAL: NCT01838551
Title: An Open Label Study to Assess the Safety and Efficacy of COR-003 (Levoketoconazole) in the Treatment of Endogenous Cushing's Syndrome
Brief Title: Treatment for Endogenous Cushing's Syndrome
Acronym: SONICS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cortendo AB (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: COR-2012-01
Record Dates: First submitted 2013-04-19; First posted 2013-04-24 (Estimated); Results first posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-03

CONDITIONS: Endogenous Cushing's Syndrome
Keywords: Cushing's disease; ectopic ACTH; adrenal Cushing's
MeSH Terms: conditions — Pituitary ACTH Hypersecretion

STUDY DESIGN:
Intervention Model Description: Dose titration
Masking Description: A data integrity plan prevented the Sponsor from accessing summary efficacy data prior to locking the clinical database.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (8):
- Levoketoconazole DL0 (Experimental): Levoketoconazole Tablets Dose Level 0 Once Daily
  Interventions: Drug: Levoketoconazole
- Levoketoconazole DL1 (Experimental): Levoketoconazole Tablets Dose Level 1 Twice Daily
  Interventions: Drug: Levoketoconazole
- Levoketoconazole DL2 (Experimental): Levoketoconazole Tablets Dose Level 1 Twice Daily
  Interventions: Drug: Levoketoconazole
- Levoketoconazole DL3 (Experimental): Levoketoconazole Tablets Dose Level 3 Twice Daily
  Interventions: Drug: Levoketoconazole
- Levoketoconazole DL4 (Experimental): Levoketoconazole Tablets Dose Level 4 Twice Daily
  Interventions: Drug: Levoketoconazole
- Levoketoconazole DL5 (Experimental): Levoketoconazole Tablets Dose Level 5 Twice Daily
  Interventions: Drug: Levoketoconazole
- Levoketoconazole DL6 (Experimental): Levoketoconazole Tablets Dose Level 6 Twice Daily
  Interventions: Drug: Levoketoconazole
- Levoketoconazole DL7 (Experimental): Levoketoconazole Tablets Dose Level 7 Twice Daily
  Interventions: Drug: Levoketoconazole

INTERVENTIONS:
Drug: Levoketoconazole — Levoketoconazole is the 2S,4R- enantiomer derived from racemic ketoconazole
  Other Names: COR-003

SUMMARY:
The primary objectives of this study are to evaluate the clinical responder rate, defined as the proportion of subjects with normal UFC after 6 months of treatment with COR-003 in the Maintenance Phase without dose increase, and to evaluate the range of effective doses in subjects with various levels of hypercortisolism.

DETAILED DESCRIPTION:
This is an open label, single arm study with a Screening Phase, a Dose Titration Phase, a 6-month Maintenance Phase, and a 6-month Extended Evaluation Phase designed to assess efficacy, safety, tolerability, and PK of COR-003 in subjects with endogenous CS.

Following an initial screening and washout period, as applicable, this study will be conducted in three treatment phases as follows:

* Dose Titration Phase: approximately 2 to 21 weeks to achieve an effective and tolerable maximum dose (the Therapeutic Dose). Dose titration will occur in increments of 150 mg with a starting dose of 150 mg twice daily (BID) over a period of approximately 2 to 21 weeks to achieve an effective and tolerable maximum dose (the Therapeutic Dose).
* Maintenance Phase: 6 months of treatment at the Therapeutic Dose following the Dose Titration Phase. Once the Therapeutic Dose has been reached and confirmed from the mean of a total of four adequately collected 24 hour urine collections for UFC measurements, subjects will enter into the Maintenance Phase of the study and will be asked to return to the clinic monthly for 6 months for assessment of efficacy and safety. During the Maintenance Phase, doses may not be increased to maintain UFC levels at or below ULN of the assay unless it is confirmed that a dose increase is deemed medically necessary at the discretion of the Investigator after discussion with the Medical Monitor. Prior to the End of Maintenance Phase Visit, four complete 24 hour urine collections will be obtained and subjects may enter the Extended Evaluation Phase.
* Extended Evaluation Phase: 6 months of continued treatment after the Maintenance Phase. In the 6-month Extended Evaluation Phase, subjects will return to the clinical site every 90 days (±14 days) for safety and efficacy evaluations.

Efficacy will be assessed primarily by measuring mean UFC concentrations at specified times as described in the clinical protocol. Safety will be assessed primarily by physical examinations with vital sign measurements, adverse events, clinical laboratory measures, electrocardiography, and pituitary MRI.

An independent Data Safety Monitoring Board (DSMB) will review the safety of the drug throughout the study. Membership of the DSMB is described in a Charter.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female ≥18 years of age
2. Able to provide written informed consent prior to any study procedures being performed; eligible subjects must be able to understand the informed consent form prior to inclusion into the study.
3. Confirmed diagnosis of newly diagnosed, persistent or recurrent Cushing's disease (CD) or endogenous CS of other etiology if subjects are not candidates for surgery or radiotherapy within the 18 months after enrollment.

   Previous medical records will be collected and used to support the diagnosis of CD or endogenous CS of other etiology, including the following etiologies:
   * Ectopic adrenocorticotropic hormone (ACTH) secretion, i.e. ACTH not of pituitary origin
   * Ectopic corticotropin-releasing hormone (CRH) secretion
   * Adrenal-dependent CS (i.e. adrenal adenoma (NOT carcinoma), adrenal hyperplasia, etc.)
   * Etiology unknown.
4. Must have elevated mean 24 hour UFC levels ≥1.5X ULN based on the normative range of the central lab assay and on a minimum of four measurements from adequately collected urine.
5. In addition to elevated mean UFC, presence of abnormal values from one of the following tests:

   * Abnormal DST: Elevated 8 AM serum cortisol ≥1.8 micrograms/dL (50 nmol/L) after 1 mg dexamethasone orally at 11 PM the evening prior (if not conducted already in the diagnostic workup of the subject within the previous 2 months before start of Screening Phase; in that case previous test results and details of conduct will need to be available by the Baseline Visit)
   * Elevated late night salivary cortisol concentrations (at least two measurements) >ULN
6. Previously irradiated subjects with CD or endogenous CS of other etiology will be allowed as long as the radiation treatment occurred > 4 years ago and subjects have not exhibited evidence for improvement in their underlying CD for 6 months prior to the Screening visit. The total number of previously irradiated subjects enrolled in this study will not exceed 10.
7. Subjects with CD or CS of other etiology who are not candidates for surgery, refuse surgery, or in whom surgery will be delayed for at least 18 months following enrollment. Subjects may be allowed to participate in the trial while awaiting surgery, but must agree to complete this study prior to surgery.
8. Subjects on treatment for CD or endogenous CS of other etiology for whom treatment has been inadequate or not well tolerated must agree to minimum washout periods prior to the Baseline Visit as specified.

Key Exclusion Criteria

1. Subjects with Pseudo-Cushing's syndrome based on assessment of the Investigator.
2. Subjects with cyclic CS based on assessment of the Investigator
3. Subjects with a non-endogenous source of hypercortisolism such as exogenous source of glucocorticoids or therapeutic use of ACTH.
4. Known inherited syndrome as the cause of hypercortisolism, including but not limited to multiple endocrine neoplasia Type 1, McCune Albright Syndrome and Carney Complex
5. Subjects with adrenal carcinoma
6. History of malignancy, other than thyroid, early stage prostate, squamous cell and basal cell carcinoma, within 3 years prior to the Screening Phase.
7. Subjects with QTc interval of >470 msec during the Screening Phase.
8. Pre-existing hepatic disease; subjects with mild to moderate hepatic steatosis consistent with fatty infiltration (non-alcoholic fatty liver disease [NAFLD] are allowed).
9. History of documented or suspected drug-induced liver injury requiring drug discontinuation of ketoconazole or any azole antifungals.
10. Subjects who receive any prohibited concomitant medication and cannot discontinue it safely prior to the Baseline Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2014-08; Primary Completion 2018-04 (Actual); Study Completion 2018-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fredric J Cohen, MD, Study Director — Cortendo AB
Locations (42):
- United States (9):
  - UCLA School of Medicine, Los Angeles, California
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - University of New Mexico HSC, Albuquerque, New Mexico
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Allegheny Neuroendocrinology Center, Pittsburgh, Pennsylvania
- University Hospitals Leuven Department of Endocrinology, Leuven, Belgium
- University Specialized Hospital for Active Treatment in Endocrinology (USHATE), Sofia, Bulgaria
- St. Pauls Hospital/Vancouver General Hospital, Vancouver, British Columbia, Canada
- Vseobecna fakultni nemocnice v Praze - III. Interni klinika VFN a 1. LF UK, Prague, Czechia
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet,Copenhagen University Hospital, Copenhagen
- Hôpital de la CONCEPTION, Service d'Endocrinologie, Diabète et Maladies Métaboliques, Marseille, France
- Med Clinic I - University of Lueback, Lübeck, Germany
- Israel (3):
  - Bnail Zion Medical Center Institute of Endocrinology & Metabolism, Haifa
  - Institute of Endocrinology & Metabolism, Rabin Medical Center, Petah Tikva
  - Sourasky Medical Center, Endocrinology & Metabolism, Tel Aviv
- Italy (9):
  - Azienda Ospedaliera-Universitaria Ancona, Ancona
  - UOC di Endocrinologia, Dipartimento di Medicina Clinica e Sperimentale, Messina
  - Istituto Auxologico Italiano, Milan
  - University of Naples Federico II, Naples
  - SCDU Medicina Interna I Università di Torino Dipartimento di Scienze Cliniche e Biologiche, Orbassano
  - University of Padua, Padua
  - Institute of Medical Pathology, Roma
  - Azienda Ospedaliero - Universitaria Città della Salute e della Scienza di Torino, Torino
  - Policlinico GB Rossi, Verona
- Netherlands (2):
  - Leiden University, Leiden University Medical Center, Dept. of Endocrinology, Leiden
  - Erasmus MC, Dpt. Of Internal Medicine, Division of Endocrinology, Rotterdam
- Poland (5):
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Terpa Sp.z.o.o, Lublin
  - Szpital Kliniczny im. Heliodora Swiecickiego, Poznan
  - Outpatient Clinic: Reuma Centrum, Warsaw
  - Samodzielny Publiczny Szpital Kliniczny Nr 1, Wroclaw
- Clinical Center of Serbia, Belgrade, Serbia
- Spain (3):
  - Hospital Universidad De La Ribera, Alzira, Valencia
  - Endocrinologia, Hospital Sant Pau,Universitat Autònoma de Barcelona, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
- Turkey (Türkiye) (2):
  - Bezmi Alem Vakıf Üniversitesi Endokrinoloji Bölümü Adnan, Istanbul
  - Istanbul University Medical Faculty, Istanbul

REFERENCES:
- [Result] Fleseriu M, Pivonello R, Elenkova A, Salvatori R, Auchus RJ, Feelders RA, Geer EB, Greenman Y, Witek P, Cohen F, Biller BMK. Efficacy and safety of levoketoconazole in the treatment of endogenous Cushing's syndrome (SONICS): a phase 3, multicentre, open-label, single-arm trial. Lancet Diabetes Endocrinol. 2019 Nov;7(11):855-865. doi: 10.1016/S2213-8587(19)30313-4. Epub 2019 Sep 18. PMID 31542384
- [Result] Geer EB, Salvatori R, Elenkova A, Fleseriu M, Pivonello R, Witek P, Feelders RA, Bex M, Borresen SW, Puglisi S, Biller BMK, Cohen F, Pecori Giraldi F. Levoketoconazole improves clinical signs and symptoms and patient-reported outcomes in patients with Cushing's syndrome. Pituitary. 2021 Feb;24(1):104-115. doi: 10.1007/s11102-020-01103-6. Epub 2020 Nov 20. PMID 33216275
- [Derived] Pivonello R, Elenkova A, Fleseriu M, Feelders RA, Witek P, Greenman Y, Geer EB, Perotti P, Saiegh L, Cohen F, Arnaldi G. Levoketoconazole in the Treatment of Patients With Cushing's Syndrome and Diabetes Mellitus: Results From the SONICS Phase 3 Study. Front Endocrinol (Lausanne). 2021 Apr 7;12:595894. doi: 10.3389/fendo.2021.595894. eCollection 2021. PMID 33897615

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Following screening, subjects were considered enrolled in the study if they met eligibility criteria, which included confirmation of increased UFC levels as per the eligibility requirements and took at least 1 dose of levoketoconazole.
Groups:
- Levoketoconazole All Doses: All doses used in the study combined
Period: Overall Study
Arm/Group | Levoketoconazole All Doses
Started | 94 (94 subjects were enrolled and received at least 1 dose of levoketoconazole)
Completed | 46 (46 subjects completed the Extended Evaluation phase)
Not Completed | 48
Not completed — Adverse Event | 16
Not completed — Death | 1
Not completed — Lack of Efficacy | 10
Not completed — Physician Decision | 4
Not completed — Withdrawal by Subject | 10
Not completed — No reason reported (2); surgery (2), cancer (1), sponsor request (1), bad clinical condition (1) | 7

BASELINE CHARACTERISTICS:
Arm/Group | Levoketoconazole All Doses
Number analyzed (Participants) | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 81
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 90
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 28
  Spain | 3
  Canada | 1
  Netherlands | 5
  Turkey | 3
  Belgium | 3
  Denmark | 4
  Poland | 8
  Italy | 20
  Israel | 9
  Bulgaria | 6
  France | 2
  Serbia | 1
  Germany | 1
Baseline 24-hour mUFC [Mean (Standard Deviation); unit: nmol/day] — Population: 2 subjects did not have sufficient adequate baseline samples for mUFC determination
  nmol/day
    number analyzed (Participants) | 92
    (all) | 671 (743)

OUTCOME MEASURES:

1. Primary Outcome: Normalization in Urinary Free Cortisol in Patients With Endogenous Cushing's Syndrome.
Description: The response to COR-003 is defined as mean UFC concentration ≤ULN following 6 months of maintenance phase therapy without a prior dose increase during that phase. The proportion of responders at the End of Maintenance Phase visit, following 6 months of treatment in the Maintenance Phase, for all dose groups combined was estimated using a generalized linear model with repeated measurements based on a binomial distribution with a logit link function and with region (US vs. non-US), concurrent CS medical conditions (diabetes [Yes/No], hypertension [Yes/No]), age (rounded median split based on the ITT population), sex, disease duration (years), prior CS medication (Yes/No), prior radiation therapy (Yes/No) as Baseline covariates and visit as an independent factor.
  The least squares mean (LSMEAN) estimate of the UFC response after 6 months of treatment in the Maintenance Phase alongside its 95% Wald CI is presented.
Time Frame: 6 months of maintenance phase therapy without a prior dose increase during that phase
Population: The primary efficacy analysis was based on the ITT population. Subjects were imputed as non-responders under any of the following conditions: withdrew anytime prior to the Month 6 of Maintenance phase; had a dose increase relative to the therapeutic dose during Maintenance phase; Month 6 mUFC data were missing or inadequate; or had received radiation therapy and exhibited no rebound increase in mUFC following withdrawal of levoketoconazole immediately after the end of Maintenance phase.
Measure: Least Squares Mean (95% Confidence Interval); unit: proportion of subjects meeting endpoint
Arm/Group | Levoketoconazole All Doses
Number analyzed (Participants) | 94
proportion of subjects meeting endpoint | .30 [.21 to .40]
Statistical Analysis 1: Comparison: Levoketoconazole All Doses; The least squares mean (LSMEAN) estimate of the UFC response after 6 months of treatment in the Maintenance Phase alongside its 95% Wald CI is presented. Supportive to the 95% CI, the p-value corresponding to the null hypothesis that the response rate is ≤ 20% is presented (1-sided test); Test type: Superiority — Under the null hypothesis of at most 20% UFC responders, 90 subjects in the ITT population would provide 90% power, with two-sided type 1 error of 0.05, assuming an observed response of 35%; p = 0.0154, Mixed Models Analysis — One-sided p-value is based on a null hypothesis that true response proportion is ≤ 0.20; The Generalized Linear Model described above was used to generate the p-value

ADVERSE EVENTS:
Time Frame: Reported adverse events are summarized for the period from the first day of study drug administration through the last day plus 30 days. For an individual subject, the maximum period of time for which adverse events were collected and summarized here (treatment-emergent only) was approximately 1 year, 11 months. For the ITT population, the median time period over which adverse events were collected and summarized was 1 year, 2 months; the mean time period was approximately 1 year.
Description: AEs were to be ascertained at each study visit by asking the subject how the subject had been since the last visit. A clinical observation, laboratory value, or imaging abnormality that the Investigator deemed clinically significant was to be recorded as an AE. An attempt was to be made to describe the AE in terms of a diagnosis. If a clear diagnosis could not be established, each sign and symptom was to be recorded individually.
Arm/Group | Levoketoconazole All Doses
All-Cause Mortality (participants affected / at risk) | 1/94
Serious Adverse Events (participants affected / at risk) | 16/94
Other Adverse Events (participants affected / at risk) | 92/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Levoketoconazole All Doses (N=94)
Pyelonephritis chronic (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Electrocardiogram QT prolonged (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Fatigue (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Benign ovarian tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Epilepsy (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Retinal artery occlusion (Eye disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Hyphaema (Injury, poisoning and procedural complications) | 1
Renal impairment (Renal and urinary disorders) | 1
Uterine polyp (Reproductive system and breast disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Levoketoconazole All Doses (N=94)
Palpitations (Cardiac disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 7
Abdominal pain upper (Gastrointestinal disorders) | 9
Diarrhea (Gastrointestinal disorders) | 14
Dyspepsia (Gastrointestinal disorders) | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 31
Vomiting (Gastrointestinal disorders) | 10
Asthenia (General disorders) | 6
Edema peripheral (General disorders) | 18
Fatigue (General disorders) | 16
Nasopharyngitis (Infections and infestations) | 12
Urinary tract infection (Infections and infestations) | 11
Alanine aminotransferase increased (Investigations) | 15
Aspartate aminotransferase increased (Investigations) | 12
Blood alkaline phosphatase increased (Investigations) | 5
Electrocardiogram QT prolonged (Investigations) | 9
Gamma-glutamyltransferase increased (Investigations) | 11
Decreased appetite (Metabolism and nutrition disorders) | 5
Hypokalemia (Metabolism and nutrition disorders) | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 14
Back pain (Musculoskeletal and connective tissue disorders) | 7
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Dizziness (Nervous system disorders) | 12
Dysgeusia (Nervous system disorders) | 6
Headache (Nervous system disorders) | 27
Anxiety (Psychiatric disorders) | 7
Insomnia (Psychiatric disorders) | 8
Menstruation irregular (Reproductive system and breast disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 9
Dry skin (Skin and subcutaneous tissue disorders) | 11
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 8
Hypertension (Vascular disorders) | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated from this study are the property of Cortendo Inc. (a subsidiary of Strongbridge Biopharma). Independent analyses and/or publication of data by Investigators is not permitted without prior written consent of Cortendo. Publication of results is to be conducted in accordance with Good Publication Practice as per Strongbridge publication policy.

DOCUMENTS (2):
  • Study Protocol (2016-10-25): https://cdn.clinicaltrials.gov/large-docs/51/NCT01838551/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-19): https://cdn.clinicaltrials.gov/large-docs/51/NCT01838551/SAP_001.pdf